CLINICAL TRIAL: NCT01235819
Title: Comparison Between GLP 1 Analogues and DPP 4 Inhibitors in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Command Hospital, India (Other Government)
Responsible Party: Principal Investigator, KVS Hari Kumar, Endocrinologist, Command Hospital, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM/CHCC/03/2010
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; exenatide; sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin; Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin alone (Active Comparator): Type 1 DM only on Insulin
  Interventions: Drug: Insulin
- Insulin and Exenatide (Active Comparator): Newly detected Type 1 DM on Insulin and exenatide
  Interventions: Drug: Exenatide
- Insulin and Sitagliptin (Active Comparator): Newly detected Type 1 DM using Insulin and Sitagliptin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Insulin — Exenatide Sitagliptin
  Other Names: Premixed Insulin
  Arms: Insulin alone
Drug: Sitagliptin — Sitagliptin 100 mg per day oral
  Other Names: DPP 4 inhibitors
  Arms: Insulin and Sitagliptin
Drug: Exenatide — Exenatide 10 micrograms daily twice
  Other Names: GLP 1 analogues
  Arms: Insulin and Exenatide

SUMMARY:
To study the effects of GLP 1 analogues and DPP 4 inhibitors on newly detected type 1 diabetes patients.

DETAILED DESCRIPTION:
Inclusion criteria T1DM <3 months GAD Antibody+ Stimulated C peptide<0.5ng/ml Ketosis at onset Age < 30 yr Exclusion criteria Age > 30 yr Pancreatic disease significant systemic complication

ELIGIBILITY:
Inclusion Criteria:

* T1DM <3 months
* GAD Antibody+ or Stimulated C peptide<0.5 ng/ml
* Ketosis at onset
* Age < 30 yr

Exclusion Criteria:

* Age > 30 yr
* Pancreas disease
* Significant systemic disease

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
change in insulin requirement | one year
  To assess the change in insulin requirement with use of GLP 1 analogues or DPP 4 inhibitors along with insulin in type 1 diabetes

SECONDARY OUTCOMES:
C peptide response | at the end of one year
  To assess the endogenous insulin secretion after one year of use of GLp 1 analogue and DPP 4 inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: The Commandant, MD, Study Director — Command Hospital
Locations (1):
- Command Hospital, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Not permitted

REFERENCES:
- [Derived] Hari Kumar KV, Shaikh A, Prusty P. Addition of exenatide or sitagliptin to insulin in new onset type 1 diabetes: a randomized, open label study. Diabetes Res Clin Pract. 2013 May;100(2):e55-8. doi: 10.1016/j.diabres.2013.01.020. Epub 2013 Mar 13. PMID 23490599